CLINICAL TRIAL: NCT00991913
Title: Risk Factors of Recovery Room Delirium After Elective Non-cardiovascular Surgery in Post-anaesthesia Care Unit
Brief Title: Risk Factors of Recovery Room Delirium After Elective Non-cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Department of Anesthesiology, Huazhong University of Science and Technology
Other Study IDs: TJHMZK02001
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Delirium
Keywords: Delirium; Postoperative; Non-cardiovascular surgery; Post-anaesthesia care unit
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Delirium: Delirium was determined by CAM-ICU
- no Delirium: no Delirium was determined by CAM-ICU

SUMMARY:
Despite recent advances in postoperative delirium research, the proportion of patients with postoperative delirium is still high ranging between 20-80%. Although postoperative delirium is a frequent complication and is associated with the need for more inpatient hospital care and longer length of hospital stay, little is known about risk factors for recovery room delirium (RRD) occurred in postanaesthesia care unit. The aim of the study was to determine pre- and intraoperative risk factors for the development of RRD among patients undergoing non cardiovascular surgery.

DETAILED DESCRIPTION:
Recovery room delirium (RRD) defined as delirium occurred in PACU was diagnosed according to CAM-ICU criteria. Pre-, intra-, and postoperative data of patients undergoing elective non cardiovascular surgery were prospectively collected, univariate and multivariate logistic regression were performed to find the risk factors related to postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiovascular surgery
* general anesthesia

Exclusion Criteria:

* under 18yr of age
* under regional anaesthesia
* refused to sign consent form
* history of substance dependence
* underwent neurosurgery
* history of primary neurologic diseases
* stayed less than 10min in PACU
* received general anaesthesia but recovered in locations outside the recovery room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18yr, who were admitted to the PACU after elective surgery under general anaesthesia during regular working hours (9:00Am to 5:00Pm)
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2010-06-01; Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of delirium in post anesthesia care unit (PACU) determined by confusion assessment method (CAM) -ICU criteria | at 1 hour after operation

SECONDARY OUTCOMES:
heart rate in PACU | every 10 mins
  heart rate was recorded every 10 min during PACU stay, maximal and minimal heart rate were collected for analysis
Pulse Oximeter Oxygen Saturation (SpO2) in PACU | every 10 mins
Hospital-length of stay | up to 6 months
Total health care fees | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China